CLINICAL TRIAL: NCT06934122
Title: Effect of Audible Manipulation Sound on Perceived Pain, Satisfaction and Disability in Non-specific Cervicothoracic Pain
Brief Title: Effect of Audible Manipulation Sound in Non-specific Cervicothoracic Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ayça Aytar (Other)
Responsible Party: Sponsor-Investigator, Ayça Aytar, Associate Professor, Baskent University
Organization: Baskent University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KA24/199
Record Dates: First submitted 2025-04-10; First posted 2025-04-18 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-05

CONDITIONS: Pain; Disability
Keywords: Neck pain; Manuel therapy
MeSH Terms: conditions — Pain; Neck Pain

STUDY DESIGN:
Intervention Model Description: To decide on the sample size, an effect size of 0.25, a Type I error of 0.05, a test power of 80% and a confidence interval of 95% were determined using the G*Power program. The first group was determined as those with an audible sound during the procedure, and the second group was determined as those with no audible sound at the end of the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- spinal manipulation (Experimental): All participants will first receive a massage and then be manipulated with the spinal manipulation technique.
  Interventions: Other: manipulation with classical massage and spinal manipulation technique

INTERVENTIONS:
Other: manipulation with classical massage and spinal manipulation technique — All participants will first receive a massage to relax the muscles and then be manipulated with a spinal manipulation technique.

SUMMARY:
The aim of this study is to investigate the effect of auditory manipulation sound on perceived pain, satisfaction and disability in patients with nonspecific cervicothoracic pain.İndividuals with nonspecific cervicothoracic pain will be included. the first group will be determined as those with an audible sound at the end of manipulation, and the second group will be determined as those without an audible sound at the end of manipulation. all evaluations and the patient's satisfaction level will be made before the application and 48 hours after the application.

DETAILED DESCRIPTION:
Before the application, the pain intensity of the individuals will be assessed with a visual analog scale, and the level of disability will be assessed with the 'neck pain and disability index'. neck mobility will be measured with a cervical inclinometer and spinal region fascia mobility modified schober test, and also the thoracolumbar fascia flexibility will be recorded. .

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of non-specific spinal pain
* Must be able to do exercise by alone

Exclusion Criteria:

* Clinical diagnosis of neurological problems (Alzheimer's, Demans)
* Clinical diagnosis of deep vein thrombosis
* Clinical diagnosis of systemic and uncontrolled metabolic diseases( Diabetes, Thyroid,hypertension)
* Don't have pain while doing exercise

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women were included to exclude the effects of different hormonal structures and gender on pain.
Enrollment: 38 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Neck mobility | immediately before starting the application and 48 hours after the application
  Neck mobility will be measured with a cervical inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: nihan özünlü pekyavaş, Principal Investigator — prof
Locations (2):
- Turkey (Türkiye) (2):
  - Başkent University, Ankara, Ankara
  - Baskent University, Ankara, Etimesgut

IPD SHARING:
Plan to Share IPD: No
We prefer to share our data and study design once they are published

REFERENCES:
- [Background] de Sousa Almeida AP, Matsui EKK, da Silva FN, de Oliveira Vasconcelos FB, de Oliveira MR. Thoracic Spine Mobility and Posture: Correlation and Predictive Values in Physically Independent Older Adults. Eval Health Prof. 2024 Mar;47(1):133-138. doi: 10.1177/01632787231220612. Epub 2023 Dec 8. PMID 38065535
- [Background] Munke Cross, P., & Ingvi Jacobsen, V. (2022). The Thrust-A Must?: a literature review of the effectiveness of thrust manipulation for pain relief in musculoskeletal conditions
- [Background] Sun X, Chai L, Huang Q, Zhou H, Liu H. Effects of exercise combined with cervicothoracic spine self-mobilization on chronic non-specific neck pain. Sci Rep. 2024 Mar 4;14(1):5298. doi: 10.1038/s41598-024-55181-8. PMID 38438448